CLINICAL TRIAL: NCT02086604
Title: A Phase I Trial of Brentuximab Vedotin in Combination With Lenalidomide in Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Brentuximab Vedotin and Lenalidomide for Relapsed or Refractory Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201404056
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Brentuximab Vedotin; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Starting Dose (brentuximab vedotin & lenalidomide) (Experimental): Brentuximab vedotin 1.2 mg/kg intravenously (IV) on Day 1 of every 21 day cycle.
  Lenalidomide 20 mg orally on Days 1-21 of every 21 day cycle.
  Interventions: Drug: Brentuximab vedotin; Drug: Lenalidomide
- Dose Level 1 (brentuximab vedotin & lenalidomide) (Experimental): Brentuximab Vedotin 1.2 mg/kg intravenously (IV) on Day 1 of every 21 day cycle.
  Lenalidomide 20 mg orally on Days 1-21 of every 21 day cycle.
  Interventions: Drug: Brentuximab vedotin; Drug: Lenalidomide
- Dose Level 2 (brentuximab vedotin & lenalidomide) (Experimental): Brentuximab Vedotin 1.2 mg/kg intravenously (IV) on Day 1 of every 21 day cycle.
  Lenalidomide 20 mg orally on Days 1-21 of every 21 day cycle.
  Interventions: Drug: Brentuximab vedotin; Drug: Lenalidomide

INTERVENTIONS:
Drug: Brentuximab vedotin
  Other Names: Adcetris®
Drug: Lenalidomide
  Other Names: Revlimid®

SUMMARY:
This Phase I clinical trial studies the side effects and maximum tolerated dose (MTD) of the combination of brentuximab vedotin (BV) and lenalidomide in the treatment of patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory de novo or transformed DLBCL disease following at least one prior systemic therapy (for DLBCL).
* CD30 immunohistochemical staining using the anti-CD30 BerH2 antibody must be available on the most recent biopsy specimen. During dose escalation, patients can be either CD30 positive or CD30 negative. During dose expansion, 15 patients must be CD30 positive and 15 patients must be CD30 negative.
* Post-ASCT or not a candidate for ASCT. Prior allogeneic stem cell transplant is allowed if patient is off all immunosuppressives and has no evidence of active GVHD.
* Prior treatment with brentuximab vedotin is allowed provided the patient did not progress on BV or within 30 days of last dose of BV. Patients must be at least 3 months from the last dose of BV.
* Bidimensional measurable disease of at least 1.5 cm in the greatest transverse diameter as documented by CT or PET/CT.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Bone marrow and organ function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1,000/mcl
  * Platelets ≥ 50,000/mcl
  * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (IULN) OR serum bilirubin ≤ 3.0 x IULN for patients with Gilbert's disease or documented hepatic involvement with NHL
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x IULN OR ALT and AST ≤ 5.0 x IULN for patients with documented hepatic involvement with NHL
  * Creatinine clearance ≥ 60 mL/min/1.73 m2 as calculated by Cockcroft-Gault
* Women of childbearing potential must follow pregnancy testing requirements as outlined in the Revlimid REMS® program material. This is defined as either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of contraception (one highly effective method and one additional effective method AT THE SAME TIME) at least 28 days prior to the start of lenalidomide, for the duration of study participation, and for 28 days following the last doses of brentuximab vedotin and lenalidomide. Women of childbearing potential must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a woman of childbearing potential even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* All study participants must be registered into the mandatory Revlimid REMS® program and be willing to comply with its requirements. Per standard Revlimid REMS® program requirements, all physicians who prescribe lenalidomide for research subjects enrolled into this trial, must be registered in, and must comply with, all requirements of the Revlimid REMS® program.
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Primary mediastinal B-cell lymphoma
* A history of other primary invasive malignancy that has not been in remission for at least 3 years or a current diagnosis of myelodysplastic syndrome (MDS) or an immature leukemia such as acute myeloid leukemia (AML).
* Known active cerebral/meningeal lymphoma.
* Present or history of progressive multifocal leukoencephalopathy (PML).
* NYHA Class III or IV congestive heart failure.
* Active CTCAE version 4.03 grade 3 or higher viral, bacterial, or fungal infection.
* Known to be positive for hepatitis B by surface antigen expression and hepatitis B core antibody.
* Known to have active hepatitis C infection (positive by polymerase chain reaction) or on antiviral therapy for hepatitis C within 6 months prior to the first doses of brentuximab vedotin and lenalidomide.
* Known to be positive for HIV.
* Receiving chemotherapy, radiotherapy, biologics, and/or other antitumor treatment with immunotherapy that is not completed at least 3 weeks prior to study entry, unless underlying disease is progressing on therapy.
* Currently receiving any other investigational agents.
* Known hypersensitivity to any excipient contained in the drug formulation of brentuximab vedotin or lenalidomide.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide.
* Receiving immunosuppressive therapy.
* Refractory to prior therapy with brentuximab vedotin (evidence of progression within 30 days of the last dose).
* Prior therapy with lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-09-18 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Safety as measured by grade and frequency of adverse events | 30 days after completion of treatment
  Adverse events will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Maximum Tolerated Dose (MTD) as measured by the number of dose-limiting toxicities in each dose level (cohort) | Completion of the first cycle for all participants in dose expansion phase (approximately 12 months)
  MTD is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle. Dose escalations will proceed until the MTD has been reached.

SECONDARY OUTCOMES:
Objective response rate as measured by CD30 expression | Up to 2 years after discontinuation of treatment
  The objective response rate by CD30 expression (proportion of positive cells, staining intensity, or both) is defined as the proportion of patients with CR or PR stratified by different values or categories of CD30 expression. Positive CD30 expression is defined as ≥1% staining of the malignant cells.
Overall response rate | Up to 2 years after discontinuation of treatment
  Complete response rate (CR) + Partial response rate (PR) = Overall response rate according to the Revised Response Criteria for Malignant Lymphoma (Cheson 2007).
Duration of response | Up to 2 years after discontinuation of treatment
  Duration of response is defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression (including radiographic and clinical progression) or to death due to any cause, whichever comes first.
  Duration of response data will be censored on the day following the date of the last disease assessment documenting absence of progressive disease for patients who do not have tumor progression and are still on study at the time of an analysis, are given antitumor treatment (including stem cell transplant) other than the study treatment, or are removed from study prior to documentation of tumor progression.
  Duration of response will only be calculated for the subgroup of patients achieving a CR or PR.
Progression-free survival (PFS) | Up to 2 years after discontinuation of treatment
  PFS is defined as the time from start of study treatment to first documentation of tumor progression (including radiographic and clinical progression) or to death due to any cause, whichever comes first.
  PFS data will be censored on the day following the date of the last disease assessment documenting absence of progressive disease for patients who do not have tumor progression and are still on study at the time of an analysis, are given antitumor treatment (including stem cell transplant) other than the study treatment, or are removed from study prior to documentation of tumor progression. Patients lacking an evaluation of tumor response after their first dose will have their event time censored at 1 day.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Bartlett, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Ohio State University, James Cancer Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ward JP, Berrien-Elliott MM, Gomez F, Luo J, Becker-Hapak M, Cashen AF, Wagner-Johnston ND, Maddocks K, Mosior M, Foster M, Krysiak K, Schmidt A, Skidmore ZL, Desai S, Watkins MP, Fischer A, Griffith M, Griffith OL, Fehniger TA, Bartlett NL. Phase 1/dose expansion trial of brentuximab vedotin and lenalidomide in relapsed or refractory diffuse large B-cell lymphoma. Blood. 2022 Mar 31;139(13):1999-2010. doi: 10.1182/blood.2021011894. PMID 34780623
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu